CLINICAL TRIAL: NCT05149430
Title: Evolution and Follow-up of the Quality of Life and Functional Capacity, in Patients Admitted in Ward Room, Post-hospitality in the Intensive Care Unit. Descriptive Study
Brief Title: Quality of Life and Functional Capacity in Post Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Sanatorio Anchorena San Martin (Other)
Collaborators: Cagide Sabrina (Unknown); Di giorgio Victoria (Unknown); Villalba Dario (Unknown); Accoce Matias (Unknown)
Responsible Party: Principal Investigator, Matias Bertozzi, Respiratory Therapy, Sanatorio Anchorena San Martin
Other Study IDs: SAnchorenaSanMartin
Record Dates: First submitted 2021-11-09; First posted 2021-12-08 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Post-intensive Care Syndrome
MeSH Terms: conditions — postintensive care syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational Quality of life and functional capacity — Observational Quality of life and functional capacity

SUMMARY:
BACKGROUND. Staying in an intensive care unit can lead to physical and cognitive complications and post-traumatic stress. Currently, the aim is to find out the level of quality of life, functional capacity and cognitive status post intensive care unit. Describe the evolution of the quality of life, functional capacity and cognitive status of a cohort of patients admitted to the ward room after discharge from the intensive care unit, with subsequent follow-up at 3, 6 and 12 months of his discharge.

METHODS. Prospective, observational, analytical cohort study. Subjects over 18 years of age with at least 48 hours of confinement in a closed area were included. Demographic variables, quality of life, functional capacity and cognitive status were recorded. A telephone follow-up was carried out three, six and twelve months after institutional discharge. For the evaluation of the primary variables, Euroqol 5d-5L (Eq5d - Eq5d-VAS), Barthel Index and Fototest were used.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years old
* At least 48 hours in the ICU
* Who subsequently entered the Clinical Ward Room
* Who signed the informed consent

Exclusion Criteria:

* Those patients who received invasive mechanical ventilation in the last 6 months
* Who had been admitted to an ICU in the last 6 months
* Patients who cannot answer the questionnaires on their own or who do not have relatives to answer them
* Patients with progressive degenerative neurological pathology.
* Patients diagnosed with cancer with a life expectancy of less than 12 months according to the criteria of the oncologist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post ICU patients who entered to the ward room
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Quality of life | 2019 - 2020
  It is the perception that an individual has of his place in existence, in the context of the culture and the value system in which he lives. This aspect was evaluated using the EuroQol Group EQ-5D-5L (EQ-5D-5L) tool.
Functional capacity | 2019 - 2020
  Functional capacity refers to the capability of performing tasks and activities that people find necessary or desirable in their lives. It was assessed using the Barthel Index (IB) tool.
Cognitive status | 2019 - 2020
  Cognitive impairment is when a person has trouble remembering, learning new things, concentrating, or making decisions that affect their everyday life.. It was evaluated by Fototest, it is a cognitive test, which includes several domains, language (denomination), executive tasks (verbal fluency) and episodic memory either free or facilitated by keys.

CONTACTS AND LOCATIONS:
Locations (1):
- Matias Bertozzi, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Needham DM, Davidson J, Cohen H, Hopkins RO, Weinert C, Wunsch H, Zawistowski C, Bemis-Dougherty A, Berney SC, Bienvenu OJ, Brady SL, Brodsky MB, Denehy L, Elliott D, Flatley C, Harabin AL, Jones C, Louis D, Meltzer W, Muldoon SR, Palmer JB, Perme C, Robinson M, Schmidt DM, Scruth E, Spill GR, Storey CP, Render M, Votto J, Harvey MA. Improving long-term outcomes after discharge from intensive care unit: report from a stakeholders' conference. Crit Care Med. 2012 Feb;40(2):502-9. doi: 10.1097/CCM.0b013e318232da75. PMID 21946660
- [Background] Herridge MS, Cheung AM, Tansey CM, Matte-Martyn A, Diaz-Granados N, Al-Saidi F, Cooper AB, Guest CB, Mazer CD, Mehta S, Stewart TE, Barr A, Cook D, Slutsky AS; Canadian Critical Care Trials Group. One-year outcomes in survivors of the acute respiratory distress syndrome. N Engl J Med. 2003 Feb 20;348(8):683-93. doi: 10.1056/NEJMoa022450. PMID 12594312
- [Background] Williams TA, Dobb GJ, Finn JC, Knuiman MW, Geelhoed E, Lee KY, Webb SA. Determinants of long-term survival after intensive care. Crit Care Med. 2008 May;36(5):1523-30. doi: 10.1097/CCM.0b013e318170a405. PMID 18434893
- [Background] Fan E, Dowdy DW, Colantuoni E, Mendez-Tellez PA, Sevransky JE, Shanholtz C, Himmelfarb CR, Desai SV, Ciesla N, Herridge MS, Pronovost PJ, Needham DM. Physical complications in acute lung injury survivors: a two-year longitudinal prospective study. Crit Care Med. 2014 Apr;42(4):849-59. doi: 10.1097/CCM.0000000000000040. PMID 24247473
- [Background] Dinglas VD, Faraone LN, Needham DM. Understanding patient-important outcomes after critical illness: a synthesis of recent qualitative, empirical, and consensus-related studies. Curr Opin Crit Care. 2018 Oct;24(5):401-409. doi: 10.1097/MCC.0000000000000533. PMID 30063492
- [Background] Spragg RG, Bernard GR, Checkley W, Curtis JR, Gajic O, Guyatt G, Hall J, Israel E, Jain M, Needham DM, Randolph AG, Rubenfeld GD, Schoenfeld D, Thompson BT, Ware LB, Young D, Harabin AL. Beyond mortality: future clinical research in acute lung injury. Am J Respir Crit Care Med. 2010 May 15;181(10):1121-7. doi: 10.1164/rccm.201001-0024WS. Epub 2010 Mar 11. PMID 20224063
- [Background] Parker A, Sricharoenchai T, Needham DM. Early Rehabilitation in the Intensive Care Unit: Preventing Physical and Mental Health Impairments. Curr Phys Med Rehabil Rep. 2013 Dec;1(4):307-314. doi: 10.1007/s40141-013-0027-9. PMID 24436844
- [Background] Steenbergen S, Rijkenberg S, Adonis T, Kroeze G, van Stijn I, Endeman H. Long-term treated intensive care patients outcomes: the one-year mortality rate, quality of life, health care use and long-term complications as reported by general practitioners. BMC Anesthesiol. 2015 Oct 12;15:142. doi: 10.1186/s12871-015-0121-x. PMID 26459381
- [Background] Rydingsward JE, Horkan CM, Mogensen KM, Quraishi SA, Amrein K, Christopher KB. Functional Status in ICU Survivors and Out of Hospital Outcomes: A Cohort Study. Crit Care Med. 2016 May;44(5):869-79. doi: 10.1097/CCM.0000000000001627. PMID 26929191
- [Background] Dettling-Ihnenfeldt DS, Wieske L, Horn J, Nollet F, van der Schaaf M. Functional Recovery in Patients With and Without Intensive Care Unit-Acquired Weakness. Am J Phys Med Rehabil. 2017 Apr;96(4):236-242. doi: 10.1097/PHM.0000000000000586. PMID 28301864
- [Background] Duarte PAD, Costa JB, Duarte ST, Taba S, Lordani CRF, Osaku EF, Costa CRLM, Miglioranza DC, Gund DP, Jorge AC. Characteristics and Outcomes of Intensive Care Unit Survivors: Experience of a Multidisciplinary Outpatient Clinic in a Teaching Hospital. Clinics (Sao Paulo). 2017 Dec;72(12):764-772. doi: 10.6061/clinics/2017(12)08. PMID 29319723
- [Background] Hermans G, Van Mechelen H, Clerckx B, Vanhullebusch T, Mesotten D, Wilmer A, Casaer MP, Meersseman P, Debaveye Y, Van Cromphaut S, Wouters PJ, Gosselink R, Van den Berghe G. Acute outcomes and 1-year mortality of intensive care unit-acquired weakness. A cohort study and propensity-matched analysis. Am J Respir Crit Care Med. 2014 Aug 15;190(4):410-20. doi: 10.1164/rccm.201312-2257OC. PMID 24825371
- [Background] Augustovski FA, Irazola VE, Velazquez AP, Gibbons L, Craig BM. Argentine valuation of the EQ-5D health states. Value Health. 2009 Jun;12(4):587-96. doi: 10.1111/j.1524-4733.2008.00468.x. Epub 2008 Nov 12. PMID 19900257
- [Background] Della Pietra GL, Savio K, Oddone E, Reggiani M, Monaco F, Leone MA. Validity and reliability of the Barthel index administered by telephone. Stroke. 2011 Jul;42(7):2077-9. doi: 10.1161/STROKEAHA.111.613521. Epub 2011 Apr 28. PMID 21527755
- [Background] Shah S, Vanclay F, Cooper B. Improving the sensitivity of the Barthel Index for stroke rehabilitation. J Clin Epidemiol. 1989;42(8):703-9. doi: 10.1016/0895-4356(89)90065-6. PMID 2760661
- [Background] Hermans G, Van den Berghe G. Clinical review: intensive care unit acquired weakness. Crit Care. 2015 Aug 5;19(1):274. doi: 10.1186/s13054-015-0993-7. PMID 26242743
- [Background] Diaz Ballve LP, Dargains N, Urrutia Inchaustegui JG, Bratos A, Milagros Percaz M, Bueno Ardariz C, Cagide S, Balestrieri C, Gamarra C, Paz D, Rotela E, Muller S, Bustos F, Aranda Castro R, Settembrino E. Weakness acquired in the intensive care unit. Incidence, risk factors and their association with inspiratory weakness. Observational cohort study. Rev Bras Ter Intensiva. 2017 Oct-Dec;29(4):466-475. doi: 10.5935/0103-507X.20170063. Epub 2017 Dec 7. PMID 29236843
- [Background] Carnero-Pardo C, Lopez-Alcalde S, Allegri RF, Russo MJ. A systematic review and meta-analysis of the diagnostic accuracy of the Phototest for cognitive impairment and dementia. Dement Neuropsychol. 2014 Apr-Jun;8(2):141-147. doi: 10.1590/S1980-57642014DN82000009. PMID 29213895
- [Background] Carnero-Pardo C, Saez-Zea C, De la Vega Cotarelo R, Gurpegui M; en nombre del grupo FOTOTRANS. [FOTOTRANS study: multicentre study on the validity of Fototest under clinical practice conditions]. Neurologia. 2012 Mar;27(2):68-75. doi: 10.1016/j.nrl.2011.06.001. Epub 2011 Sep 1. Spanish. PMID 21889232
- [Background] Sacanella E, Perez-Castejon JM, Nicolas JM, Masanes F, Navarro M, Castro P, Lopez-Soto A. Functional status and quality of life 12 months after discharge from a medical ICU in healthy elderly patients: a prospective observational study. Crit Care. 2011;15(2):R105. doi: 10.1186/cc10121. Epub 2011 Mar 28. PMID 21443796
- [Background] Pintado MC, Villa P, Lujan J, Trascasa M, Molina R, Gonzalez-Garcia N, de Pablo R. Mortality and functional status at one-year of follow-up in elderly patients with prolonged ICU stay. Med Intensiva. 2016 Jun-Jul;40(5):289-97. doi: 10.1016/j.medin.2015.08.002. Epub 2015 Dec 23. English, Spanish. PMID 26706825
- [Background] Hopkins RO, Miller RR 3rd, Rodriguez L, Spuhler V, Thomsen GE. Physical therapy on the wards after early physical activity and mobility in the intensive care unit. Phys Ther. 2012 Dec;92(12):1518-23. doi: 10.2522/ptj.20110446. Epub 2012 Apr 5. PMID 22491481
- [Background] Rollinson TC, Connolly B, Berlowitz DJ, Berney S. Physical activity of patients with critical illness undergoing rehabilitation in intensive care and on the acute ward: An observational cohort study. Aust Crit Care. 2022 Jul;35(4):362-368. doi: 10.1016/j.aucc.2021.06.005. Epub 2021 Aug 10. PMID 34389239
- [Background] Griffiths J, Hatch RA, Bishop J, Morgan K, Jenkinson C, Cuthbertson BH, Brett SJ. An exploration of social and economic outcome and associated health-related quality of life after critical illness in general intensive care unit survivors: a 12-month follow-up study. Crit Care. 2013 May 28;17(3):R100. doi: 10.1186/cc12745. PMID 23714692
- [Background] Herridge MS, Tansey CM, Matte A, Tomlinson G, Diaz-Granados N, Cooper A, Guest CB, Mazer CD, Mehta S, Stewart TE, Kudlow P, Cook D, Slutsky AS, Cheung AM; Canadian Critical Care Trials Group. Functional disability 5 years after acute respiratory distress syndrome. N Engl J Med. 2011 Apr 7;364(14):1293-304. doi: 10.1056/NEJMoa1011802. PMID 21470008
- [Background] Brower RG. Consequences of bed rest. Crit Care Med. 2009 Oct;37(10 Suppl):S422-8. doi: 10.1097/CCM.0b013e3181b6e30a. PMID 20046130
- [Background] Linko R, Suojaranta-Ylinen R, Karlsson S, Ruokonen E, Varpula T, Pettila V; FINNALI study investigators. One-year mortality, quality of life and predicted life-time cost-utility in critically ill patients with acute respiratory failure. Crit Care. 2010;14(2):R60. doi: 10.1186/cc8957. Epub 2010 Apr 12. PMID 20384998
- [Background] Eggmann S, Luder G, Verra ML, Irincheeva I, Bastiaenen CHG, Jakob SM. Functional ability and quality of life in critical illness survivors with intensive care unit acquired weakness: A secondary analysis of a randomised controlled trial. PLoS One. 2020 Mar 4;15(3):e0229725. doi: 10.1371/journal.pone.0229725. eCollection 2020. PMID 32131082
- [Background] Das Neves AV, Vasquez DN, Loudet CI, Intile D, Saenz MG, Marchena C, Gonzalez AL, Moreira J, Reina R, Estenssoro E. Symptom burden and health-related quality of life among intensive care unit survivors in Argentina: A prospective cohort study. J Crit Care. 2015 Oct;30(5):1049-54. doi: 10.1016/j.jcrc.2015.05.021. Epub 2015 Jun 3. PMID 26105747
- See also: Related Info — https://scirp.org/reference/referencespapers.aspx?referenceid=1138949
- See also: Das Neves A, Busico M, Yanes N. Síndrome post terapia intensiva. Evaluación, prevención y seguimiento. En: Programa de actualización en kinesiología intensivista (PROAKI), ciclo 2, módulo 4. Editorial Médica Panamericana. Vol. 4. 2015. — http://revista.ajrpt.com/index.php/Main/article/view/88
- See also: Related Info — https://clincalc.com/IcuMortality/Default.aspx
- See also: Related Info — http://www.scielo.org.ar/scielo.php?script=sci_arttext&pid=S1852-236X2014000300008

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT05149430/SAP_000.pdf